CLINICAL TRIAL: NCT05856422
Title: Respiratory Rate Validation Study - Gabi SmartCare Gabi Band
Brief Title: Respiratory Rate Validation Study
Status: Completed | Type: Interventional
Sponsor: Gabi SmartCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RR3
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Measure Accuracy of Respiratory Rate
Keywords: respiratory rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Pediatrics population (Experimental)
  Interventions: Device: Respiratory rate measure based on PPG

INTERVENTIONS:
Device: Respiratory rate measure based on PPG — Testing was conducted under normal office environment conditions. Each subject was connected to the reference EtCO2 monitor (GE Datex-Ohmeda) and the Device Under Test, the Gabi SmartCare Gabi Band. A waveform collected from an EtCO2 measurement was used to determine performance of respiratory rate metrics. Each subject was given a nasal cannula that allowed for measurement of the EtCO2 respiratory rate.
  The reference respiratory rate was measured simultaneously with the Device Under Test. Data was marked for stable quiet periods that were useable for analysis.

SUMMARY:
The purpose of this study is to conduct a Respiratory Rate accuracy validation on pediatrics population comparing the Gabi SmartCare Gabi Band to the Reference, an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex- Ohmeda) by manually scoring the collected waveform for data analysis.

DETAILED DESCRIPTION:
Each participant is expected to take 1-2 hours, including paperwork, sensor application, and a maximum of 60 minutes of data collection. Each participant will be connected to a commonly used End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda) and the Gabi SmartCare Gabi Band. The end tidal carbon dioxide (EtCO2) monitor will determine performance of respiratory rate metrics (GE Healthcare S5 Compact Monitor with M-COVX (K001814) or E-CaiO (K051092) modules). Each participant will be instrumented with neonatal or pediatric nasal cannula that allows for measurement of the EtCO2. SpO2 sensors may be placed on the feet and/or toes for safety monitoring purposes.

Data will be simultaneously and continuously recorded from the Reference EtCO2 monitor and the Device Under Test (DUT). Periods of quiet will be encouraged. Data will be marked for stable quiet periods that are useable for analysis. There is no additional follow-up required for the investigation.

One minute epochs will be generated from the stable data periods for analysis. For verification, the Reference EtCO2 waveform will be scored by counting the respiratory peaks per minute.

The reviewers counting the raw EtCO2 waveform will be blinded to the results from the test device. The DUT data will be averaged over the corresponding one minute period. The Accuracy root- mean-square (Arms) will be the basis for evaluation and acceptance.

To 'Pass' this test the Gabi SmartCare Gabi Band (Device Under Test) must demonstrate an Accuracy root-mean- square (Arms) of ≤3.0 breaths per minute when compared to the Reference EtCO2 monitor.

The study population will include a minimum of 23 neonates, infants, and pediatrics from 0-12 years of age. A maximum of 60 participants will be enrolled. The participant selection will be an equitable distribution of males and females of any race with varying skin tones. An attempt will be made to include 3 darkly pigmented participants (Fitzpatrick 5 or 6) or 15% of the participant pool (whichever is larger).

The parents or guardian of the participants must understand the study and consent to their child's participation in the study by signing the Informed Consent Form. Subjects 7 to 12 years of age will be provided an Assent. The study will be explained within his/her ability to understand. Participant enrollment and participation in this clinical study is based on meeting the inclusion criteria and none of the exclusion criteria, a satisfactory screening, and the participant and data demographics needed for the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability of the parent or guardian to understand and provide written informed consent
* Participant is 0 to 12 years of age
* Subjects that are between 7 and 12 years of age must provide Assent to participate in the study

Exclusion Criteria:

* Participants evaluated by the Investigator and Clinical Staff and found to be medically unsuitable or have self-reported health conditions that are currently unstable as identified in the Participant Demographics and Screening Record Form
* Participant has injuries, deformities or abnormalities that may prevent proper application of the device under test
* Participants with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, or other medical sensors (self-reported)

Ages: 1 Minute to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark LLC, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pediatrics Population
Started | 21
Completed | 13
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pediatrics Population
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Device Under Test for the Measurement of Respiratory Rate, Measured in Breath/Min
Description: Arms or rms error, given in breath per minute, is the calculation of root mean square between Respiratory rate of the subject device and the manually scored reference Respiratory Rate EtCO2 waveform, for all stable respiratory periods. It is a way of averaging the absolute values of errors over the full measurement range and is a similar measurement to a "rms error". It indicates how far (accurate) the provided value is from the reference used. A passing result required an Arms of ≤3 breaths/min.
Time Frame: Every 60 seconds, over a total duration of maximum 60 minutes
Measure: Number; unit: breaths/min
Arm/Group | Pediatrics Population
Number analyzed (Participants) | 13
breaths/min | 2.9

ADVERSE EVENTS:
Time Frame: During the period of measurement and 15 minutes after, up to 75 minutes
Arm/Group | Pediatrics Population
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT05856422/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT05856422/SAP_001.pdf